CLINICAL TRIAL: NCT02167568
Title: Corpus Callosum Agenesis and Intellectual Disability: Genetic and Phenotypic Characterization
Brief Title: Corpus Callosum Agenesis and Intellectual Disability
Acronym: ACCREM
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P081260
Record Dates: First submitted 2014-06-13; First posted 2014-06-19 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-06

CONDITIONS: Intellectual Deficiency; Cerebral Abnormality
Keywords: corpus callosum agenesis/dysgenesis; mental deficiency/ Intellectual deficiency; genetic and phenotypic characterization
MeSH Terms: conditions — Agenesis of Corpus Callosum; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Corpus callosum agenesis/dysgenesis: patients with Corpus callosum agenesis/dysgenesis
  Interventions: Genetic: Genetic
- parents: parents of patients with corpus callosum agenesis/dysgenesis
  Interventions: Genetic: Genetic

INTERVENTIONS:
Genetic: Genetic

SUMMARY:
Corpus callosum agenesis or dysgenesis (CCA) is a major brain malformation (˜1/4000 births) presently diagnosed by prenatal ultrasonography. In about half of the cases, CCA is associated with other anomalies (complex CCA), which usually leads to medical abortion. Syndromes including a CCA are many (hundreds), most of which are also associated with intellectual deficiency (ID). Several genes are involved in such complex CCA. On the other hand, several studies pointed to the favorable cognitive outcome of individuals/fetuses with an apparently isolated CCA (ICCA) during pregnancy in about 70% of cases. However, there are still 30% of cases with ID or developmental delay. The precise incidence and severity of these disorders are presently unclear. Therefore, prenatal counseling of couples facing a prenatal diagnosis of ICCA is still elusive.

Our aims are to unravel the genetic causes of CCA by combining phenotypic and genetic analyses in a prospective cohort of patients with CCA and intellectual disability, in order to improve prenatal information.

DETAILED DESCRIPTION:
Corpus callosum is the main midline brain structure connecting homologous cortical areas of both hemispheres. Corpus callosum agenesis or dysgenesis (CCA) can be diagnosed antenatally, either isolated or associated with other cerebral or extra-cerebral malformations. With an incidence of 1.8/10,000 newborn, CCA is often associated with chromosomal anomalies and mendelian syndromes. Even when CCA appears to be isolated, the neuro-developmental outcome is uncertain, with many children developing normally, and others having moderate learning disabilities or even severe ID. The genetic heterogeneity of complex CCA is large (CCA can be observed in more than 300 entities), but for many patients, no etiological diagnosis is known. Therefore, genetic counselling remains challenging in many cases. Recurrence is observed in almost 5% of cases, and for most patients with no etiological diagnosis, the disease is sporadic. These data suggest both recessive and dominant de novo inheritance.

This study aims, in a prospective cohort of 120 patients with CCA and intellectual disability:

1. To determine the nature and the frequency of characterized genetic abnormalities.
2. To determine the phenotypic spectrum of complex CCA
3. To perform SNP-array analyses (i) for patients without etiological diagnosis and (ii) for patients with an identified syndrome without molecular basis to clarify the genetic basis of CCA and to evaluate the contribution of this technique in these patients
4. To describe new clinical- genetic entities

Patients are recruited through pediatric neurology and genetics consultations in the reference and competence centers " intellectual disabilities of rare cause" and associated network called "DéfiSciences".

The workup will include for all patients :

1. a clinical examination by a neurologist and a clinical geneticist, and a child psychiatric care if needed
2. a blood sample for patient and his parents 2.3. a neuropsychological assessment if needed 3.4. Cerebral MRI using new technologies (diffusion, tracking fiber spectroscopy ... ) , if not available Central reviews of brain MRI are performed by a referent neuroradiologist in order to classify the type of CCA, morphological features and associated brain abnormalities.

4.5. Several additional tests could be performed if necessary:

a. in search of associated malformations i. renal ultrasound ii. echocardiogram iii. bone x-rays iv. ophthalmological examination b. in search of neurological/sensorial dysfunction: neurophysiological assessment (electroencephalogram, brainstem evoked auditory potentials, somatosensory evoked potentials, electroretinogram and visual evoked potentials) c. Karyotype d. Molecular biology: ARX(for boys) XFRA e. Metabolic tests comprising at least plasma CK, chromatography of plasma amino acids, chromatography of urine organic acids, a redox cycle, urinary creatine and guanidinoacetic acid assay and a Bratton-Marshall test ;

After this initial assessment, investigators of the core clinical/research team will discuss all cases to validate proposed diagnoses and to determine whether a secondary assessment or complementary genetic studies are needed. Patients without established diagnosis will benefit from a study using whole genome chips (Illumina SNP-array) to be conducted at the end of the recruitment period for the second year of the project. This work will improve the essential clinical and genetic knowledge of CCA, which is necessary to improve the assessment of the prognosis in prenatal diagnosis and genetic counseling. It is also expected to expand the understanding of the complex development of the corpus callosum and its function.

ELIGIBILITY:
Inclusion criteria :

* age > 3 months
* patient with mental retardation
* patient with corpus callosum agenesis (complete or partial) or dysgenesis

Exclusion criteria :

* Patient with corpus callosum agenesis or dysgenesis but without mental retardation
* Patient with mental retardation but with total callosum corpus(cc)
* Patient with corpus callosum agenesis or dysgenesis and mental retardation whose origin is acquired
* Patient does not wish to participate, or whose parents / guardians refuse their participation
* Patient in whom brain MRI cannot be performed
* Patient not affiliated to a social security system (or beneficiaries who right) or CMU
* Patient with at least one of the two parent's inclusion it not possible

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patient with corpus callosum agenesis (complete or partial) or dysgenesis associated to mental retardation recruted through pediatric neurology and genetics consultations in the reference and competence centers " intellectual disabilities of rare cause" and associated network called "DéfiSciences".
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2012-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
genetic abnormalities | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Delphine HERON, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Groupe Hospitalier Pitié-Salpêtrière, Paris, France